CLINICAL TRIAL: NCT00511576
Title: A Phase 1, Open-Label, Dose-Escalation Trial to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of MGCD0103 (MG-0103) in Combination With Docetaxel (Taxotere®) in Subjects With Advanced Solid Malignancies
Brief Title: Study to Evaluate Combination Treatment of MGCD0103 and Docetaxel (Taxotere®) for Subjects With Advanced Cancer Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Celgene terminated its collaboration agreement with MethylGene for the development of MGCD0103. All Celgene-sponsored trials with MGCD0103 will be closed.
Sponsor: Mirati Therapeutics Inc. (Industry)
Responsible Party: Gregory Reid, Executive Director, Clinical Development, MethylGene Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 103 PH US 2007 CL001
Record Dates: First submitted 2007-08-03; First posted 2007-08-06 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2015-01

CONDITIONS: Breast Cancer; Lung Cancer; Pulmonary Cancer; Non-Small-Cell Lung Carcinoma; Prostate Cancer; Prostatic Cancer; Gastric Cancer; Stomach Cancer
Keywords: Advanced or Metastatic Breast Cancer; Breast Cancer; Advanced or Metastatic Non-Small-Cell Lung Cancer (NSCLC); Hormone Refractory Prostate Cancer; Prostate Cancer; Gastric Cancer; Advanced Gastric Adenocarcinoma; HDAC Inhibitor; Taxotere; Docetaxel
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Prostatic Neoplasms; Stomach Neoplasms | interventions — mocetinostat; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part 1 (Active Comparator): In Part 1, cohorts of three to six subjects will receive doses of MGCD0103 administered orally three times per week (TIW) in combination with 60 mg/m2 IV docetaxel administered as a 1-hour infusion on Day 1 of each 3-week (21-day) cycle. The starting dose of MGCD0103 in Part 1 will be 50 mg (approximately 25 mg/m2).
  Interventions: Drug: MGCD0103 & Docetaxel
- Part 2 (Active Comparator): Part 2 will begin once the MTD for MGCD0103 in combination with 60 mg/m2 IV docetaxel has been determined and further evaluated in the expansion phase. In Part 2, cohorts of three to six subjects will receive escalating doses of MGCD0103 administered orally TIW in combination with 75 mg/m2 docetaxel administered as a 1-hour IV infusion on Day 1 of each cycle. The starting dose of MGCD0103 administered in combination with 75 mg/m2 IV docetaxel will be the MTD from Part 1 minus 25 mg.
  Interventions: Drug: MGCD0103 & Docetaxel

INTERVENTIONS:
Drug: MGCD0103 & Docetaxel — In both Parts 1 and 2, subsequent doses of MGCD0103 will be escalated in 25 mg increments until the MTD of MGCD0103 in combination with each fixed dose (60 mg/m2 or 75 mg/m2) ofIV docetaxel is determined.
  In both parts 1 and 2, MGCD0103 will be administered orally TIW for 3 weeks beginning on Day 1 at 1 hour prior to the start of the IV docetaxel infusion.
  There will be no scheduled break between cycles and no limit to the number of cycles a subject can receive provided they do not have disease progression as defined by RECIST, or a clinically significant drug-related adverse event (AE) that does not resolve or respond to treatment intervention with 3 weeks.
  Other Names: MG-0103; Taxotere®

SUMMARY:
The purpose of this study is to test the combination of an experimental drug known as MGCD0103 given along with an FDA-approved drug called docetaxel. This is a Phase 1 study that will look at different doses of MGCD0103 given along with docetaxel in order to better understand the effects (positive and negative) of this combination on the subject's body and disease.

The study would like to find the following information:

* How long MGCD0103 and docetaxel stay in the subject's body;
* What effects, good and/or bad, MGCD0103 and docetaxel have on the subject and on his/her cancer; and
* If the genetic and chemical make-up of the subject's blood cells and tumor cells play a role in how you respond or do not respond to MGCD0103 and docetaxel.

DETAILED DESCRIPTION:
This Phase 1 study will evaluate escalating doses of orally administered MGCD0103 in combination with two fixed doses (60 mg/m2 and 75 mg/m2) of IV docetaxel. In the US, docetaxel is recommended at these or even higher doses (up to 100 mg/m2), both as a single agent or in combination with other cytotoxic drugs (e.g., cisplatin, doxorubicin, cyclophosphamide, and 5-fluorouracil), for the treatment of NSCLC, prostate cancer, gastric adenocarcinoma, and head and neck cancer. In Japan, 60 mg/m2 IV docetaxel is the approved dose for the treatment of breast cancer.

MGCD0103 belongs to the class of more selective, less globally cytotoxic agents being investigated for treatment of cancers today, and may offer a lesser and/or non-overlapping toxicity profile than the cytotoxic agents with which docetaxel is currently combined. MGCD0103 doses ranging from 50 to 135 mg have been administered in combination with the approved regimen of azacitidine (Vidaza®) (75 mg/m2/day for 5 days every 4 weeks) to patients with high-risk MDS and AML. A 50 mg dose of MGCD0103 has been administered in combination with the approved regimen of gemcitabine (1000 mg/m2 once weekly for 3 consecutive weeks of each 4-week cycle) to patients with advanced solid tumors; higher doses of MGCD0103 will soon be evaluated in that trial.

Given the above, the proposed starting dose of 60 mg/m2 IV docetaxel and 50 mg MGCD0103 is considered appropriately safe for initial investigation of this combination. Based on the results observed in Part 1, the study may also evaluate 75 mg/m2 IV docetaxel and escalating doses of orally administered MGCD0103 in Part 2 in order to determine whether this dosing regimen is safe and would also warrant further investigation.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet ALL inclusion criteria to be enrolled in the study

* Age ≥18 years.
* Diagnosis of malignant solid tumor (histologically or cytologically confirmed) where treatment with docetaxel is considered standard of care, or advanced solid malignancy that has failed to respond to standard therapy, or has progressed despite standard therapy, or where there is no reasonable likelihood of achieving clinical benefit with existing therapies.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2.
* Adequate organ function, including: Hemoglobin (Hgb) ≥8.0g/dL; Absolute neutrophil count (ANC) ≥1.5 x 10<9>/L (≥1500/mm<3>); Platelets ≥100 x 10<9>/L (≥100,000/mm<3>); Total bilirubin ≤1.5 x ULN (upper limit of normal); AST (SGOT) and ALT (SGPT) ≤2.5 x ULN; Alkaline phosphatase ≤5.0 x ULN; Serum creatinine ≤2.0 x ULN.
* Evidence of measurable disease (ie, at least one lesion that can accurately be measured in at least one dimension as ≥20 mm with conventional techniques or ≥10 mm with spiral CT scan). The requirement for measurable disease will not apply to subjects with prostate cancer.
* A minimum of 4 weeks elapsed since any major surgery.
* At least 4 weeks elapsed since any prior anticancer therapy (standard or investigational) and full recovery (NCI CTCAE grade 1) from the toxic effects of that treatment. Antiandrogen therapy is permitted for subjects with prostate cancer.
* For women of childbearing potential, a negative serum pregnancy test within 10 days of treatment, and use of physician-approved methods of birth control throughout the study.
* Written, informed consent, willingness, and ability to comply with all study procedures.

Exclusion Criteria:

Subjects meeting any of the following criteria will not be included in the study.

* Prior taxane and HDAC inhibitor combination therapy.
* Previous or concurrent malignancy except adequately treated basal cell or squamous cell skin cancer; in situ carcinoma of the cervix, or other solid tumor treated curatively, and without evidence of recurrence for at least 3 years prior to study entry.
* Clinically significant cardiac disease including congestive heart failure (New York Heart Association Class III or IV), including pre-existing ventricular arrhythmia or conduction abnormality requiring medication, or cardiomyopathy.
* Active and uncontrolled clinically significant infection.
* History of melena, hematemesis, or hemoptysis within the last 3 months.
* Known central nervous system metastases controlled ≤3 months.
* Pregnant or lactating women. Women of child-bearing potential must have a negative serum pregnancy test within 10 days of starting study drug on Day 1 Cycle 1.
* Known hypersensitivity to taxanes, HDAC inhibitors, and/or any components of MGCD0103 capsules or docetaxel formulation components (eg, polysorbate 80).
* Known HIV or known active Hepatitis B or C.
* Presence of serious illness, medical condition, or other medical history, including abnormal laboratory parameters, which, in the opinion of the Investigator, would be likely to interfere with a subject's participation in the study or with the interpretation of the results.
* Any condition that will put the subject at undue risk or discomfort as a result of adherence to study procedures (eg, requirement to take MGCD0103 with a low pH beverage).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2007-08; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD), dose limiting toxicities (DLTs), and safety profile of escalating doses of orally administered MGCD0103 in combination with two fixed doses (60 mg/m2 and 75 mg/m2) of IV docetaxel. | 15 months
To assess the plasma pharmacokinetics (PK) of MGCD0103 (and/or its metabolites) and IV docetaxel administered in combination. | 15 months
To evaluate potential pharmacodynamic (PD) effects of orally administered MGCD0103 in combination with IV docetaxel. | 15 months
To determine the overall tumor response of orally administered MGCD0103 in combination with IV docetaxel according to Response Evaluation Criteria in Solid Tumors (RECIST) methodology. | 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Reid, MSc, MBA, Study Director — MethylGene Inc.
Locations (2):
- United States (2):
  - Johns Hopkins, Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - University of Pennsylvania, Philadelphia, Pennsylvania